CLINICAL TRIAL: NCT06442163
Title: Outcome Measures of Auto-titrating Average Volume-assured Pressure Support (AVAPS) as Rescue Therapy After CPAP Titration Failure in Patients With Obesity Hypoventilation Syndrome: Adherence and Sleep Quality
Brief Title: Average Volume-assured Pressure Support as Rescue Therapy in Obesity Hypoventilation Syndrome
Acronym: AVAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Magdy Eid, professor of pulmonary medecine, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5000231
Record Dates: First submitted 2024-05-18; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
Keywords: ventilation, Obesity
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Respiratory Aspiration; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Clinically stable OHS patients with a body mass index of 30 kg/m2 and daytime hypercapnia (PaCO2 (Experimental): Each participant underwent initial baseline diagnostic polysomnograms (PSG) documenting the presence of OSA based on standard diagnostic criteria. After baseline (PSG) and patient's consent, patients performed full night CPAP titration in the sleep laboratory within 7 days of the baseline PSG, and AVAPS-AE titration.
  Interventions: Device: AVAPS study was performed within 1 week of the CPAP titration attempt failure, using the auto-titrating EPAP (AE), the OmniLab Advanced +, System One device (Philips Respironics, Murrysville, PA, U.S.

INTERVENTIONS:
Device: AVAPS study was performed within 1 week of the CPAP titration attempt failure, using the auto-titrating EPAP (AE), the OmniLab Advanced +, System One device (Philips Respironics, Murrysville, PA, U.S. — After attending an educational session (in the presence of a family member) with hands-on training, the AVAP -AE devices were provided to the patients.
  During the study, one month after AVAPS -AE initiation, patients had direct immediate access to medical and technical support through phone contact during daytime working hours.

SUMMARY:
It remains unclear whether CPAP therapy should be prescribed if significant hypoxemia persists during CPAP titration, despite optimization of upper airway obstructive events, if maximum CPAP pressure is reached.

The goal was to examine the effects of 6 months of home AVAPS therapy in patients with obesity hypoventilation syndrome as a potential option for patients who failed CPAP titration due to persistent hypoxemia.

DETAILED DESCRIPTION:
Obesity hypoventilation syndrome (OHS) is one of the leading indications of home non-invasive ventilation (NIV) initiation. In patients with OHS, NIV improves daytime vigilance, decreases PaCO2, improves sleep quality, and improves physical activity.

Thus, the primary aim of this study was to evaluate the effects of 6-month noninvasive ventilation with average volume-assured pressure support (AVAPS-AE) ventilation on objective sleep quality and adherence to therapy in stable patients with OHS who failed CPAP titration.

ELIGIBILITY:
Inclusion Criteria:

* All Clinically stable OHS patients with

  * Body mass index of 30 kg/m2 ,
  * Daytime hypercapnia (PaCO2 >45 mm Hg) who had failed to respond to CPAP therapy
  * had no other cause for their chronic respiratory failure and were naive to any PAP therapy.

Exclusion Criteria:

* Patients with evidence of acute respiratory failure (patients with worsening symptoms during the last 2 weeks before the screening visit, a breathing frequency of 30 breaths/ minute, or signs of respiratory infections)
* Patients who had been intubated during the last 3 months
* Patients who had received any other form of ventilatory support before hospital admission were also excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
To compare the initial diagnostic, and therapeutic sleep study parameters using either CPAP and (AVAPS-AE) titration study in patients with OHS. | 1 week
  polysomnographic parameter (apnea hypopnea index (events/hours)

SECONDARY OUTCOMES:
The effects of 6 month of home AVAPS- AE therapy on patient adherence and sleep quality in OHS patients who failed CPAP titration due to persistent hypoxemia. | at 1 ,3,6 months
  Patients had follow-up appointments at two distinct time points, after 3 month and final visit after 6 month of home AVAPS- AE therapy, to address sleep quality using: Self-assessed sleep quality (0: very poor/10: very good). Objective assessment of adherence to AVAPS- AE therapy was recorded. The ATS criteria defined "good adherence" to PAP as "using PAP therapy regularly for > 4 h/night for >70% of the recorded time"

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Magdy, Principal Investigator — Assiut University
Locations (1):
- Assuit University Hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No
after being published